CLINICAL TRIAL: NCT00626821
Title: An Open Label, Non-comparative, Multi-national Post-Market Study to Document Real Life Experience on SenSura With Focus on Skin Condition and Quality of Life
Brief Title: Coloplast DialogueStudy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK175OS
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Results first posted 2012-03-12 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-01

CONDITIONS: Stoma
Keywords: Stoma; Ostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: SenSura

INTERVENTIONS:
Device: SenSura — Real life assessment of SenSura

SUMMARY:
The main purpose of the study is to document real life experience on SenSura with focus on skin condition and quality of life.

DETAILED DESCRIPTION:
It is important to continuously develop and test ostomy products in order to prevent peristomal skin disorders and to enhance the quality of life for people with a stoma. Furthermore, it is essential to create awareness about the importance of healthy peristomal skin as many of these conditions are preventable.

ELIGIBILITY:
Inclusion criteria

* Signed informed consent before any study related activities
* Subjects with a colostomy, ileostomy or urostomy
* Subjects must have had their ostomy for at least 6 months
* Subjects must have mental capacity to understand the study and questionnaires
* Subjects must be at least 18 years of age.

Exclusion criteria

* Women who are pregnant or breast-feeding
* Subjects who have more than one ostomy
* Subjects with an ostomy who use plug
* Participation in other studies at the same time
* Previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3017 (Actual)
Dates: Start 2008-02; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte D Andersen, RN, Principal Investigator — Herlev Hospital, Dep of colorectal surgery
Locations (1):
- Restored Images, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SenSura: Test of SenSura for 6-8 weeks
Period: Overall Study
Arm/Group | SenSura
Started | 3017
Quality of Life | 2672 (Attended both visit 1 and visit 2)
Completed | 2796
Not Completed | 221
Not completed — Adverse Event | 44
Not completed — Protocol Violation | 33
Not completed — Withdrawal by Subject | 10
Not completed — Physician Decision | 9
Not completed — Product dysfunction | 21
Not completed — other/unknown reason | 104

BASELINE CHARACTERISTICS:
Arm/Group | SenSura
Number analyzed (Participants) | 3017
Age Continuous [Mean (Standard Deviation); unit: years] | 63.2 (14.3)
Gender [Number; unit: participants] — Gender is unknown for 2 participants
  participants
    Female | 1541
    Male | 1474

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life (Scale 0(Worst)-100(Best))
Description: The mean change in quality of life (Stoma-QoL value) from visit 1 to visit 2. An increase in Stoma-QoL is an improvement, a decrease in Stoma-QoL is a worsening.
Time Frame: 6-8 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- SenSura: Participants tested SenSura for 6-8 weeks. Baseline data were informations about pre-study product.
Arm/Group | SenSura
Number analyzed (Participants) | 2672
units on a scale | 1.8 (6.9)
Statistical Analysis 1: Comparison: SenSura; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 1.813, 95% CI 2-sided [1.553 to 2.073], Standard Error of Mean 0.133

ADVERSE EVENTS:
Arm/Group | SenSura
Serious Adverse Events (participants affected / at risk) | 17/3017
Other Adverse Events (participants affected / at risk) | 58/3017
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SenSura (N=3017)
Fistula surgery (Surgical and medical procedures) | 1 (1)
Scar infection (Infections and infestations) | 1 (1)
(General disorders) | 1 (1) — Only the outcome, death, has been registered
Short bowel syndrome (Gastrointestinal disorders) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 1 (1)
Surgery for ruptured disc (Surgical and medical procedures) | 1 (1)
Food blokage in the bowel (Gastrointestinal disorders) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Bowel perforation (Injury, poisoning and procedural complications) | 1 (1)
Placement of nephrostomal cathether (Surgical and medical procedures) | 1 (1)
Exhaustion (General disorders) | 1 (1) — Due to chemotherapy
Apoplexia (Nervous system disorders) | 1 (1)
Cardio respiratory arrest (Cardiac disorders) | 1 (1) — Outcome: death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SenSura (N=3017)
Peristomal skin disorder (Skin and subcutaneous tissue disorders) | 52 (52)
Gastrointeritis (Gastrointestinal disorders) | 2 (2)
(General disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less